CLINICAL TRIAL: NCT03663543
Title: The Use of Peri-Operative Intravenous Estrogen for the Mitigation of Ischemia Reperfusion Injury in the Setting of Renal Transplantation
Brief Title: Intravenous Estrogen in Kidney Transplant Study
Acronym: PERT
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 82378
Record Dates: First submitted 2018-08-27; First posted 2018-09-10 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Ischemia Reperfusion Injury
MeSH Terms: conditions — Reperfusion Injury | interventions — Estrogens, Conjugated (USP); Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Parallel: Participants are assigned to one of two or more groups in parallel for the duration of the study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Arm (Active Comparator): Participants randomized to the active arm will receive a single infusion of conjugated estrogens at the time of admission if within 8 hours of the expected surgery time or at approximately 8 hours to the expected surgery time if admission is earlier than that. Participants will then receive two daily infusions of conjugated estrogens after transplant given at 8 hours after reperfusion of the transplanted kidney and 24 hours after the first post transplant dose (32 hours after reperfusion of the transplanted kidney).
  Interventions: Drug: Conjugated Estrogen
- Placebo Arm (Placebo Comparator): Participants randomized to the placebo arm will receive normal saline (0.9% sodium chloride) at the same rate as the active arm.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Conjugated Estrogen — Dosing of conjugated estrogen will be given pre kidney transplant procedure and twice after reperfusion of the transplanted kidney.
  Other Names: Premarin
  Arms: Active Arm
Drug: Normal saline — Dosing of normal saline will be given pre kidney transplant procedure and twice after reperfusion of the transplanted kidney.
  Other Names: 0.9% sodium chloride
  Arms: Placebo Arm

SUMMARY:
Ischemia perfusion injury (IRI) is a major cause of organ injury during kidney transplantation. Currently there are no treatments for IRI other than dialysis. Preliminary studies in female mice have found protection from IRI when given short term estrogen supplements. This study will look at the effect of intravenous estrogen given peri-operatively to reduce the effect of IRI in female kidney transplant recipients.

DETAILED DESCRIPTION:
Ischemia-reperfusion injury (IRI) is a major etiology of organ injury and dysfunction that occurs during transplantation. In renal transplantation, the clinical manifestation of IRI is delayed graft function (DGF), typically defined as a recipient requiring dialysis within the first week after transplant. At present, there are no directed treatments for IRI associated with kidney transplantation and resultant DGF, other than supportive care with dialysis. This represents an unmet clinical need. While dialysis enables the support of patients until DGF resolves, DGF is associated with increased medical costs, increased length of hospital stay, increased rates of readmission to the hospital after transplantation, increased rates of rejection, and decreased graft survival. Therapies to reduce IRI might alleviate clinical complications associated with DGF, reduce costs associated with transplantation, and ease organ shortages by facilitating use of more marginal organs.

Despite acceptance of gender disparities in IRI tolerance in animal systems, attempts to utilize hormonal manipulation in humans to achieve improved IRI tolerance have not been undertaken. In an effort to design such a translation, the investigators investigated if similar gender disparities exist in humans who have undergone kidney transplantation. After review of the United Network for Organ Sharing database, the investigators established that male recipient gender was highly associated with DGF. Then, the investigators demonstrated that manipulation of the pre-ischemic environment with short-term estrogen supplementation in female mice provides protection from renal IRI. As a logical next stop, the investigators propose hormonal manipulation with perioperative administration of intravenous conjugated estrogens as a novel therapeutic strategy to reduce the effect of IRI in female humans undergoing kidney transplantation. The investigators have designed an investigational new drug (IND) late phase I/early phase II prospective, single center, double blind, randomized, placebo-controlled trial to test the safety, feasibility, and efficacy of this therapy. If the administration of peri-operative intravenous administration has a positive impact on the rate of recovery of GFR after renal transplant and the inherent IRI, then this therapy would represent the first treatment for IRI and ultimately might reduce the incidence of DGF. Because DGF after kidney transplantation is associated with inferior transplant outcomes and increased costs,2 a therapy that mitigates the effect of IRI and consequently reduces the incidence of DGF not only might alleviate these complications but could also ease organ shortages by facilitating the use of more marginal organs. Moreover, if estrogen therapy does mitigate IRI in the setting of renal transplantation, it could be applied to other causes of renal IRI including supra-celiac clamping in trauma or vascular surgery or the use of cardiopulmonary bypass in cardiac surgery. Female adult subjects with a diagnosis of end stage renal disease who are dialysis dependent at the time of deceased donor renal transplantation and meet the inclusion and exclusion criteria will be eligible for participation in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Female gender
2. Age > 21 years at time of transplant
3. Pre-existing dialysis dependence of at least 1-months duration at the time of transplant
4. Receiving a deceased donor renal transplant with KDPI >40
5. Written informed consent obtained from subject and ability for subject to comply with the requirements of the study

Exclusion Criteria:

1. History of solid organ transplant
2. Receiving a combined heart-kidney transplant, liver-kidney transplant, or other multi-visceral organ transplant
3. Personal history of deep vein thrombosis (DVT) or pulmonary embolism (PE)
4. Personal history of hypercoagulable condition including but not limited to Lupus Anticoagulant, Leiden Factor V Mutation, Prothrombin Gene Mutation, Protein C or S deficiency, or any other hypercoagulable condition considered by the attending transplant surgeon on clinical service or Data and Safety Monitoring Board (DSMB) to warrant exclusion from the study
5. Personal history of an estrogen sensitive cancer (breast, endometrial, ovarian)
6. Personal history of arterial thromboembolic disease such as stroke or myocardial infarction in the 6 months prior to transplantation
7. Patient already on estrogen (including oral contraceptive pills) or anti-estrogen therapy for other indications
8. Patient who is expected to not tolerate a dose of 500-5000U intravenous heparin at the time of transplant as determined by the transplant surgeon
9. Patient who has a contraindication or allergy to or is expected to not tolerate a dose of 2500-7500U subcutaneous heparin prophylaxis three times daily during hospital stay as determined by the transplant surgeon
10. Pregnant and breast feeding patients will be excluded from the study due to the small risk of radiation associated with the DTPA renal scan
11. Patient body mass index (BMI) > 40
12. Known anaphylactic reaction and/or angioedema to Premarin Intravenous therapy
13. Presence of a condition or abnormality that in the opinion of the investigator or attending transplant surgeon primarily responsible for the patient's care would compromise the safety of the patient or the quality of the data.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must be female
Enrollment: 30 (Estimated)
Dates: Start 2016-08-26 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Glomerular filtration rate (GFR) | Post-operative day three
  GFR (glomerular filtration rate) as calculated from a DTPA (Diethylenetriamine Pentaacetic Acid, a medication) renal scan.

SECONDARY OUTCOMES:
Delayed graft function (DGF) | Immediately post-operative
  Measurement of urine creatinine clearance and serum creatinine.

OTHER OUTCOMES:
Graft Failure | Post-operative day three and day ninety
  Measurement of serum creatinine.
Post Op Day 3 Creatinine | Post-operative day 3
  Measurement of serum creatinine and percent change from pre-transplant creatinine
Nadir Post op Day 90 Creatinine | post transplant day 90
  Measurement of serum creatinine and percent change from pre-transplant creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Levine, MD, PhD, Principal Investigator — University of Pennsylvania Health System
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siedlecki A, Irish W, Brennan DC. Delayed graft function in the kidney transplant. Am J Transplant. 2011 Nov;11(11):2279-96. doi: 10.1111/j.1600-6143.2011.03754.x. Epub 2011 Sep 19. PMID 21929642
- [Background] Kher A, Meldrum KK, Wang M, Tsai BM, Pitcher JM, Meldrum DR. Cellular and molecular mechanisms of sex differences in renal ischemia-reperfusion injury. Cardiovasc Res. 2005 Sep 1;67(4):594-603. doi: 10.1016/j.cardiores.2005.05.005. PMID 15950202
- [Background] Kher A, Wang M, Tsai BM, Pitcher JM, Greenbaum ES, Nagy RD, Patel KM, Wairiuko GM, Markel TA, Meldrum DR. Sex differences in the myocardial inflammatory response to acute injury. Shock. 2005 Jan;23(1):1-10. doi: 10.1097/01.shk.0000148055.12387.15. PMID 15614124
- [Background] Hedges SJ, Dehoney SB, Hooper JS, Amanzadeh J, Busti AJ. Evidence-based treatment recommendations for uremic bleeding. Nat Clin Pract Nephrol. 2007 Mar;3(3):138-53. doi: 10.1038/ncpneph0421. PMID 17322926
- [Background] Wigginton JG, Pepe PE, Idris AH. Rationale for routine and immediate administration of intravenous estrogen for all critically ill and injured patients. Crit Care Med. 2010 Oct;38(10 Suppl):S620-9. doi: 10.1097/CCM.0b013e3181f243a9. PMID 21164406
- [Background] Bradley LD, Gueye NA. The medical management of abnormal uterine bleeding in reproductive-aged women. Am J Obstet Gynecol. 2016 Jan;214(1):31-44. doi: 10.1016/j.ajog.2015.07.044. Epub 2015 Aug 5. PMID 26254516
- [Background] Murray AW, Barnfield MC, Waller ML, Telford T, Peters AM. Assessment of glomerular filtration rate measurement with plasma sampling: a technical review. J Nucl Med Technol. 2013 Jun;41(2):67-75. doi: 10.2967/jnmt.113.121004. Epub 2013 May 8. PMID 23658207
- [Result] Ojo AO, Wolfe RA, Held PJ, Port FK, Schmouder RL. Delayed graft function: risk factors and implications for renal allograft survival. Transplantation. 1997 Apr 15;63(7):968-74. doi: 10.1097/00007890-199704150-00011. PMID 9112349
- [Result] Alves MG, Oliveira PJ, Carvalho RA. Substrate selection in hearts subjected to ischemia/reperfusion: role of cardioplegic solutions and gender. NMR Biomed. 2011 Nov;24(9):1029-37. doi: 10.1002/nbm.1640. Epub 2011 Jan 28. PMID 21274961
- [Result] Ardelt AA, Carpenter RS, Lobo MR, Zeng H, Solanki RB, Zhang A, Kulesza P, Pike MM. Estradiol modulates post-ischemic cerebral vascular remodeling and improves long-term functional outcome in a rat model of stroke. Brain Res. 2012 Jun 21;1461:76-86. doi: 10.1016/j.brainres.2012.04.024. Epub 2012 Apr 21. PMID 22572084
- [Result] Eckhoff DE, Bilbao G, Frenette L, Thompson JA, Contreras JL. 17-Beta-estradiol protects the liver against warm ischemia/reperfusion injury and is associated with increased serum nitric oxide and decreased tumor necrosis factor-alpha. Surgery. 2002 Aug;132(2):302-9. doi: 10.1067/msy.2002.125718. PMID 12219027
- [Result] Gabel SA, Walker VR, London RE, Steenbergen C, Korach KS, Murphy E. Estrogen receptor beta mediates gender differences in ischemia/reperfusion injury. J Mol Cell Cardiol. 2005 Feb;38(2):289-97. doi: 10.1016/j.yjmcc.2004.11.013. Epub 2005 Jan 20. PMID 15698835
- [Result] Peng X, Wang J, Lassance-Soares RM, Najafi AH, Sood S, Aghili N, Alderman LO, Panza JA, Faber JE, Wang S, Epstein SE, Burnett MS. Gender differences affect blood flow recovery in a mouse model of hindlimb ischemia. Am J Physiol Heart Circ Physiol. 2011 Jun;300(6):H2027-34. doi: 10.1152/ajpheart.00004.2011. Epub 2011 Mar 11. PMID 21398592
- [Result] Hu H, Wang G, Batteux F, Nicco C. Gender differences in the susceptibility to renal ischemia-reperfusion injury in BALB/c mice. Tohoku J Exp Med. 2009 Aug;218(4):325-9. doi: 10.1620/tjem.218.325. PMID 19638737
- [Result] Muller V, Szabo A, Viklicky O, Gaul I, Portl S, Philipp T, Heemann UW. Sex hormones and gender-related differences: their influence on chronic renal allograft rejection. Kidney Int. 1999 May;55(5):2011-20. doi: 10.1046/j.1523-1755.1999.00441.x. PMID 10231466
- [Result] Muller V, Losonczy G, Heemann U, Vannay A, Fekete A, Reusz G, Tulassay T, Szabo AJ. Sexual dimorphism in renal ischemia-reperfusion injury in rats: possible role of endothelin. Kidney Int. 2002 Oct;62(4):1364-71. doi: 10.1111/j.1523-1755.2002.kid590.x. PMID 12234307
- [Result] Park KM, Kim JI, Ahn Y, Bonventre AJ, Bonventre JV. Testosterone is responsible for enhanced susceptibility of males to ischemic renal injury. J Biol Chem. 2004 Dec 10;279(50):52282-92. doi: 10.1074/jbc.M407629200. Epub 2004 Sep 8. PMID 15358759
- [Result] Park KM, Cho HJ, Bonventre JV. Orchiectomy reduces susceptibility to renal ischemic injury: a role for heat shock proteins. Biochem Biophys Res Commun. 2005 Mar 4;328(1):312-7. doi: 10.1016/j.bbrc.2004.12.177. PMID 15670785
- [Result] Robert R, Ghazali DA, Favreau F, Mauco G, Hauet T, Goujon JM. Gender difference and sex hormone production in rodent renal ischemia reperfusion injury and repair. J Inflamm (Lond). 2011 Jun 9;8:14. doi: 10.1186/1476-9255-8-14. PMID 21658244
- [Result] Rusai K, Prokai A, Szebeni B, Meszaros K, Fekete A, Szalay B, Vannay A, Degrell P, Muller V, Tulassay T, Szabo AJ. Gender differences in serum and glucocorticoid regulated kinase-1 (SGK-1) expression during renal ischemia/reperfusion injury. Cell Physiol Biochem. 2011;27(6):727-38. doi: 10.1159/000330081. Epub 2011 Jun 17. PMID 21691090
- [Result] Shen SQ, Zhang Y, Xiong CL. The protective effects of 17beta-estradiol on hepatic ischemia-reperfusion injury in rat model, associated with regulation of heat-shock protein expression. J Surg Res. 2007 Jun 1;140(1):67-76. doi: 10.1016/j.jss.2006.10.022. Epub 2007 Mar 2. PMID 17336333
- [Result] Soljancic A, Ruiz AL, Chandrashekar K, Maranon R, Liu R, Reckelhoff JF, Juncos LA. Protective role of testosterone in ischemia-reperfusion-induced acute kidney injury. Am J Physiol Regul Integr Comp Physiol. 2013 Jun 1;304(11):R951-8. doi: 10.1152/ajpregu.00360.2012. Epub 2013 Apr 3. PMID 23552495
- [Result] Wittnich C, Belanger MP, Askin N, Boscarino C, Wallen WJ. Lower liver transplant success in females: gender differences in metabolic response to global ischemia. Transplant Proc. 2004 Jun;36(5):1485-8. doi: 10.1016/j.transproceed.2004.05.055. PMID 15251365
- [Result] Antus B, Liu S, Yao Y, Zou H, Song E, Lutz J, Heemann U. Effects of progesterone and selective oestrogen receptor modulators on chronic allograft nephropathy in rats. Nephrol Dial Transplant. 2005 Feb;20(2):329-35. doi: 10.1093/ndt/gfh602. Epub 2004 Dec 23. PMID 15618244
- [Result] Antus B, Yao Y, Song E, Liu S, Lutz J, Heemann U. Opposite effects of testosterone and estrogens on chronic allograft nephropathy. Transpl Int. 2002 Oct;15(9-10):494-501. doi: 10.1007/s00147-002-0449-2. Epub 2002 Sep 20. PMID 12389082
- [Result] Aufhauser DD Jr, Wang Z, Murken DR, Bhatti TR, Wang Y, Ge G, Redfield RR 3rd, Abt PL, Wang L, Svoronos N, Thomasson A, Reese PP, Hancock WW, Levine MH. Improved renal ischemia tolerance in females influences kidney transplantation outcomes. J Clin Invest. 2016 May 2;126(5):1968-77. doi: 10.1172/JCI84712. Epub 2016 Apr 18. PMID 27088798
- [Result] Livio M, Mannucci PM, Vigano G, Mingardi G, Lombardi R, Mecca G, Remuzzi G. Conjugated estrogens for the management of bleeding associated with renal failure. N Engl J Med. 1986 Sep 18;315(12):731-5. doi: 10.1056/NEJM198609183151204. PMID 3018561
- [Result] Heistinger M, Stockenhuber F, Schneider B, Pabinger I, Brenner B, Wagner B, Balcke P, Lechner K, Kyrle PA. Effect of conjugated estrogens on platelet function and prostacyclin generation in CRF. Kidney Int. 1990 Dec;38(6):1181-6. doi: 10.1038/ki.1990.331. PMID 1963650
- [Result] Vigano G, Gaspari F, Locatelli M, Pusineri F, Bonati M, Remuzzi G. Dose-effect and pharmacokinetics of estrogens given to correct bleeding time in uremia. Kidney Int. 1988 Dec;34(6):853-8. doi: 10.1038/ki.1988.260. PMID 2850395
- [Result] DeVore GR, Owens O, Kase N. Use of intravenous Premarin in the treatment of dysfunctional uterine bleeding--a double-blind randomized control study. Obstet Gynecol. 1982 Mar;59(3):285-91. PMID 6281704